CLINICAL TRIAL: NCT07384182
Title: Assessment of Clinical and Refractive Outcomes of the Use of a Femtosecond to Treat the Symptoms of Presbyopia in a Patient With Implanted Mono Focal IOLs
Brief Title: Clinical Outcomes of Femtosecond Laser Presbyopia Treatment in Monofocal IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perfect Lens, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL-RISO1
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (1):
- Application of Perfector laser treatment (Experimental): Active treatment arm
  Interventions: Device: Perfector

INTERVENTIONS:
Device: Perfector — The Perfector is used in the procedure. The Device is attached to the patient by the use of a patient attachment. The patient attachment attaches to the sclera of the eye using vacuum pressure.

SUMMARY:
This study aimed to assess the safety and efficacy of treating presbyopia in eyes implanted with a mono focal IOL using a low-energy femtosecond laser.

DETAILED DESCRIPTION:
An investigative device built by Perfect Lens was used to adjust an implanted IOL in 38 eyes.

The device uses a femtosecond laser, a scanner, and an OCT. Each patient was presbyopic pre-treatment. The primary endpoint for the treatment was to create near vision in the treated eye without sacrificing the existing far vision. The first patient was treated in October 2023 and the last patient was treated in July 2024. The last patient visit was in November 2024.

The patients were examined at 7 days, 30 days and 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand study requirements, follow study instructions and to return for required study follow-up visits as confirmed by provision of written informed consent;
2. Subject has undergone cataract surgery and has had a monofocal lens implanted in both eyes;
3. Subject has no significant residual visual issues which the Investigator believes would make the patient ill suited for the Treatment.; and
4. Both eyes have CDVA vision of 20/25 or better at 4m.

Exclusion Criteria:

1. Subjects not able to complete the informed consent form;
2. Clinically significant corneal abnormalities including corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy), inflammation, keratitis, keratoconjunctivitis, keratouveitis, keratopathy, keratectasia or edema per the Investigator's expert medical opinion;
3. Previous corneal surgery;
4. Previous refractive surgery or proposed refractive surgery procedures throughout the entire duration of the subjects' participation in the clinical study (including, but not limited to LASIK, astigmatic keratotomy and limbal relaxing incisions);
5. History of or current retinal conditions or predisposition to retinal conditions including retinal detachment, diabetic retinopathy, age related macular degeneration which are assessed to by investigator to confound outcomes;
6. Amblyopia;
7. History of or current anterior or posterior segment inflammation of any etiology, or any disease-producing an inflammatory reaction in the eye (e.g., iritis or uveitis);
8. Optic nerve atrophy;
9. Iris neovascularization;
10. Subjects with diagnosed degenerative eye disorders (e.g., macular degeneration or other retinal disorders);
11. Uncontrolled glaucoma;
12. Any subject currently participating in another investigational drug or device studies; and
13. Any subject disqualified by the Principal Investigator or Medical Monitor for any ocular issue.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Distance corrected near visual acuity (DCNVA) at 40 cm | 1 month after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using the manifest refraction and the hand-held, 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 40 centimeters (cm) on the nearpoint rod. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
  The hypothesis tested for is to demonstrate superiority of the near vision of treated IOL to the IOL pre-treatment.
Distance corrected intermediate visual acuity (DCIVA) at 66 cm | 1 month after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using the manifest refraction and the hand-held, 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 66 centimeters (cm) on the nearpoint rod. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
  The hypothesis tested for is to demonstrate non-inferiority of the treated IOL to the pre-treated IOL (using a non-inferiority margin of 0.10 logMAR).
Corrected distance visual acuity (CDVA) at 4 m | 1 month after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using the manifest refraction adjusted for infinity and stand Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 4 meters (m) on the nearpoint rod. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
  The hypothesis tested for the co-primary effectiveness endpoint is to demonstrate non-inferiority of the treated IOL to the pre-treatment IOL (using a non-inferiority margin of 0.10 logMAR).

SECONDARY OUTCOMES:
Uncorrected distance visual acuity (UDVA) | 1 week, 1month and 3 months after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) adjusted for infinity and stand Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 4 meters (m) on the nearpoint rod. Without the manifest refraction. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Uncorrected intermediate visual acuity at 66 cm (UIVA) | 1 week, 1month and 3 months after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 66 centimeters (cm) on the nearpoint rod. Without manifest refraction. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Uncorrected near visual acuity at 40 cm (UNVA) | 1 week, 1month and 3 months after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 40 centimeters (cm) on the nearpoint rod. Without manifest refraction. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Corrected near visual acuity at 40 cm (CNVA) | 1 week, 1month and 3 months after treatment
  Visual acuity (VA) was tested monocularly and binocularly (both eyes together) using manifest refraction100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 40 centimeters (cm) on the nearpoint rod. VA was measured in logarithm minimum angle of resolution (logMAR) increments, with 0.1 logMAR corresponding to 5 letters, or 1 line, on the ETDRS chart. A lower logMAR value denotes better visual acuity.
Defocus curve | 1month and 3 months after treatment
  To assess the defocus curve the same optotype as for the distance visual acuity will be used. The test will be performed with the best distance corrected refraction and spherical additions between -5.0 D to +1.5 D in 0.5 D steps. Defocus curve will be performed monocularly. The patient will be presented with the spherical additions in the order from -5.0 D to +1.5 D.
Contrast sensitivity | 3 months after treatment
  Contrast sensitivity testing will be performed monocularly with the distance-corrected study eye under photopic with glare, mesopic and mesopic with glare conditions using CSV 1000. The testing will be performed at spatial frequencies of 3, 6, and 12 and 18 cycles/degree.
  Mesopic contrast sensitivity testing (3 cd/m2) using mesopic filter installed in the patient trial frame, will be performed prior to the photopic testing (85 cd/m2). A minimum of 5 minutes should be provided for the patient's eye dark adaptation before the beginning of the mesopic contrast testing in a room with photopic light conditions.
  The ambient illumination should be lower or at most equal to the chart luminance. The mesopic testing without glare will be performed first before testing with glare source provided with the testing device
Subjective refraction | 1 week, 1month and 3 months after treatment
  The assessment of refraction, which includes sphere (D), cylinder (D), and axis (°), will be conducted through subjective and objective methods. Objective refraction will follow standard clinical practice and will be performed by the Investigator or trained staff. Subjective testing will be conducted using trial frames instead of a phoropter. Consistency in the refractive technique should be maintained throughout the entire study duration. Test optotypes such as Sloan letters (e.g., ETDRS charts) will be used.
  The cylinder value should be recorded in negative notation. Cylinder refraction should be performed for every patient. If the cylinder refraction is zero, the cylinder axis should be marked as not applicable. A pre-sign for the sphere is only necessary for negative values. If no pre-sign is entered, it indicates a positive value
Near addition | 1 week, 1 month and 3 months after treatment
  Monocular CNVA with near addition. Designed to create additional foci in the implanted IOL which will give near vision without loss of far vision.
Slit Lamp examination findings | 1 week, 1month and 3 months after treatment
  Slit lamp examination will be performed using a slit lamp biomicroscope. The subject will be seated. During this examination the eyes might be dilated depending on doctors' decision. The following will be examined during the examination conjunctiva, cornea, anterior chamber, iris, eyelid. Magnification will be consistent with standard clinical practise.
  The observation will be graded as normal or abnormal. In case of abnormal observations subjective graded according to the grading scales will be used. The abnormal grading will then be graded as clinical significant or not clinically significant. In case of clinically significant observation the event will be specified and will be collected as adverse events.
Fundus examination findings | 1 week, 1month and 3 months after treatment
  To examine the retinal integrity and document the safety of the procedure a full fundus examination will be performed using a slit lamp and dilated pupil for a clear view.
Intraocular pressure | 1 week, 1month and 3 months after treatment
  The intraocular pressure (IOP) will be measured using air tonometry
Spectacle independence questionnaire | 3 months after treatment
  The questionnaire in the Czech language will be explained to the patient and handed over by the staff. It consists of 9 questions with multiple-choice answers as standard.
  The questions request answers on the following scale: All the time / Most of the time / Sometimes / Rarely / Never.
  The best response is never.
QoV patient questionnaire | 3 months after treatment
  The questionnaire in the Czech language will be explained to the patient and handed over by the staff. It consists of 10 questions as standard. All of the questions have 4 possible answers: Never / Occasionally / Often / Frequently. The worst outcome is frequently.
Adverse Events | 1 week, 1month and 3 months after treatment
  During the course of the planned clinical investigation, utmost attention will be given to detecting any potential adverse events or unfavourable discoveries.All findings related to adverse events must be documented in the "Adverse Event (AE)" section of the subject's worksheets (CRFs). These events are categorized as either serious or non-serious, as well as related or unrelated to the investigational device/procedure. The method of reporting or documenting these adverse events varies depending on their category (serious or non-serious).
Device deficiency | 1 week, 1 month and 3 months after treatment
  An inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety usability, safety or performance. Device deficiencies include includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling. This definition includes device deficiencies related to the investigational medical device. DD can become (might lead to) serious adverse events (SAE) if:
  1. suitable action had not been taken, or
  2. intervention had not been made, or
  3. if circumstances had been less fortunate These DDs are handled using the SAE reporting system.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, PhD FEBOS-CR, Principal Investigator — Gemini Eye Center
Locations (1):
- Gemini Eye Clinic, Zlín, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The individual participant data will be shared upon release of the Clinical Study Report. No end date.
Access Criteria: Access will be available for analysis for any purpose.

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT07384182/Prot_000.pdf
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT07384182/ICF_001.pdf